CLINICAL TRIAL: NCT05063032
Title: Left Atrial FLUTter: a Comparison of Ablation Guided by High-density MApping and Empirical LINEar Ablation - the FLUTMALINE Trial
Brief Title: Left Atrial FLUTter: a Comparison of Ablation Guided by High-density MApping and Empirical LINEar Ablation.
Acronym: FLUTMALINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Dr. Sergio Castrejón-Castrejón, Electrophysiologist, Principal investigator (togheter with Dr. José Luis Merino), Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5825 v 3.0, 3030th March 2021
Record Dates: First submitted 2021-09-07; First posted 2021-09-30 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Arrhythmias, Cardiac
Keywords: Left atrial flutter; Linear ablation; High-density mapping
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: 1:1 parallell, randomized, controlled, open-label, single center clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-density mapping guided ablation (Experimental): High-density map and return-cycles map in order to localize the protected isthmus with precision for focal/minimal ablation.
  Interventions: Other: Radiofrecuency ablation
- Empirical linear ablation (Active Comparator): Empirical predefined set of linear ablation.
  Interventions: Other: Radiofrecuency ablation

INTERVENTIONS:
Other: Radiofrecuency ablation — Radiofrequency ablation to treat left atrial flutter, guided by high-density mapping versus linear ablation.

SUMMARY:
Unicenter, 1:1 randomized, open-labelled clinical trial comparing left atrial flutter ablation using high density mapping or strict lineal ablation. Main outcome: arrhythmia recurrences over 1 year follow-up with daily 1-lead 30 seconds ECG samples.

ELIGIBILITY:
Inclusion criteria

* Left atrial flutter1 inducible during electrophysiological evaluation.
* Clinical indication for ablation: a) symptoms (palpitations, dizziness, syncope, breathlessness, derangement, heart failure), tachymiopathy, b) poor heart rate control, or c) recurrence after electrical cardioversion or failure of one antiarrhythmic drug.
* Informed consent.

  1. Patients will be enrolled if LAFL is clinically suspected but finally randomized if this mechanism is established by electrophysiologic evaluation according to the criteria stated above.

Exclusion criteria

* Previous ablation of LAFL.
* Previous linear ablation in the LA except for pulmonary vein isolation.
* Absolute contraindication for oral anticoagulation.
* Stroke or acute coronary syndrome less than 3 months before ablation.
* Complex congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients without sustained (≥30 s) atrial arrhythmia episodes over 1-year follow-up in each group. | 1 year follow-up
  Daily 1-lead 30 seconds ECG samples.

SECONDARY OUTCOMES:
Acute success. | Acute intraprocedural.
  Termination of all organized atrial arrhythmias (spontaneous or induced, organized and stable atrial arrhythmias with duration ≥3 min).
Non-inducibility. | Acute intraprocedural.
  Non-inducibility of all organized atrial arrhythmias at the end of the ablation procedure.
Procedure duration. | Acute intraprocedural.
  From vein puncture up to seaths withdrawal.
Left atrial dwell time. | Acute intraprocedural.
  From transeptal puncture up to catheters withdrawal from the left atrium.
Safety. | Acute a 1 month after ablation (procedure-related complications).
  Incidence of compications: 1)vascular lesions, 2)cardiac tamponade, 3)embolism.
Hospitalization. | 1 year.
  Number of hospitalizations due to atrial arrhythmia episodes at 1-year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Department of Cardiology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No